CLINICAL TRIAL: NCT00193297
Title: A Phase II Study of a Three-Day Schedule of Topotecan Plus Paclitaxel and Carboplatin on Day Three in the Initial Treatment of Advanced Ovarian and Primary Peritoneal Carcinoma
Brief Title: Topotecan Plus Paclitaxel and Carboplatin in the Initial Treatment of Advanced Ovarian and Primary Peritoneal Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: SCRI Oncology Research Consortium, SCRI
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI GYN 08; 104864-644
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2011-05-03 (Estimated); Status verified 2011-05

CONDITIONS: Ovary Cancer
Keywords: Ovary Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Topotecan; Paclitaxel; Carboplatin

INTERVENTIONS:
Drug: Topotecan
Drug: Paclitaxel
Drug: Carboplatin

SUMMARY:
The purpose of this study is to evaluate the feasibility and toxicity of the combination of paclitaxel, carboplatin, and topotecan in patients with previously untreated, stage III or IV epithelial ovarian carcinoma or primary peritoneal carcinoma. We will also make a preliminary evaluation of the efficacy of this three drug regimen in the initial treatment of these patients.

DETAILED DESCRIPTION:
Upon determination of eligibility, all patients will be receive:

Paclitaxel + Carboplatin + Topotecan

a maximum of six courses of chemotherapy will be given at 21 day intervals

ELIGIBILITY:
Inclusion Criteria:

To be included in this study, you must meet the following criteria:

* Epithelial ovarian carcinoma or primary peritoneal carcinoma
* Willing to consider second-look surgery to evaluate response if necessary
* No previous treatment with chemotherapy or radiation therapy
* Ability to perform activities of daily living with minimal assistance
* Adequate bone marrow, liver and kidney function
* Written informed consent

Exclusion Criteria:

You cannot participate in this study if any of the following apply to you:

* Age < 18 years
* Brain metastases
* Recent history of significant heart disease within 6 months
* Other significant medical conditions

Please note: There are additional inclusion/exclusion criteria. The study center will determine if you meet all of the criteria. If you do not qualify for the trial, study personnel will explain the reasons. If you do qualify, study personnel will explain the trial in detail and answer any questions you may have.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2002-02; Primary Completion 2005-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Overall response rate

SECONDARY OUTCOMES:
Overall toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Greco, MD, Principal Investigator — SCRI Development Innovations, LLC